CLINICAL TRIAL: NCT03077854
Title: A Single-Blind Randomized Trial of Image-Guided Functional Lung Avoidance Thoracic Radiotherapy for Locally Advanced Non-Small Cell and Small Cell Lung Cancer
Brief Title: Image-Guided Functional Lung Avoidance Thoracic Radiotherapy for Lung Cancer: A Single-Blind Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201604007RINA
Record Dates: First submitted 2016-06-27; First posted 2017-03-13 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Small Cell Lung Cancer, Limited Stage; Stage III Non-small Cell Lung Cancer
Keywords: Lung Cancer; Radiotherapy; Biomarkers; Radiation Lung Injury; Quality of Life
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Functional Lung Avoidance-TRT (Experimental): Functional Lung Avoidance Thoracic Radiotherapy
  The avoidance thoracic radiotherapy treatment plan will be designed to optimize such that radiation dose to functional lung identified by four-dimensional (4D) CT ventilation imaging is as low as reasonably achievable
  Interventions: Radiation: Functional Lung Avoidance Thoracic Radiotherapy
- Standard-TRT (Active Comparator): Standard Thoracic Radiotherapy
  The standard thoracic radiotherapy treatment plan will be designed without reference to the functional lung 4D CT ventilation imaging
  Interventions: Radiation: Standard Thoracic Radiotherapy

INTERVENTIONS:
Radiation: Functional Lung Avoidance Thoracic Radiotherapy — * Chemoradiation for non-small cell lung cancer: 60 Gy in 30 once-daily fractions (Dose reduction to 54 Gy in 30 once-daily fractions is allowed)
  * Radiation alone for non-small cell lung cancer: 60 Gy in 25 once-daily fractions (Dose reduction to 55 Gy in 25 once-daily fractions is allowed)
  * Chemoradiation for small-cell lung cancer: 45 Gy in 30 twice-daily fractions
  Arms: Functional Lung Avoidance-TRT
Radiation: Standard Thoracic Radiotherapy — * Chemoradiation for non-small cell lung cancer: 60 Gy in 30 once-daily fractions (Dose reduction to 54 Gy in 30 once-daily fractions is allowed)
  * Radiation alone for non-small cell lung cancer: 60 Gy in 25 once-daily fractions (Dose reduction to 55 Gy in 25 once-daily fractions is allowed)
  * Chemoradiation for small-cell lung cancer: 45 Gy in 30 twice-daily fractions
  Arms: Standard-TRT

SUMMARY:
Thoracic radiotherapy (TRT) is a standard curative treatment for locally advanced, unresectable non-small cell lung cancer (NSCLC) and limited stage small cell lung cancer (SCLC). TRT has been recognized to cause moderate to severe lung injury in a substantial portion of patients. Conventional standard curative TRT planning techniques minimize the radiation dose to the anatomical lungs, without adaption of regional pulmonary function variations. The principal investigator hypothesized that preferential avoidance of functional lung during curative TRT may decrease the risk of pulmonary toxicity. Functional lung regions are identified using four- dimensional computed tomography for ventilation imaging. This randomized, single-blind trial will comprehensively assess the impact of functional lung avoidance on pulmonary toxicity, quality of life, and clinical outcome in patients receiving curative TRT for locally advanced NSCLC and SCLC.

ELIGIBILITY:
Inclusion criteria:

1. Patients with a histologic diagnosis of non-small cell carcinoma or small cell carcinoma of lung
2. Locally advanced stage III A or III B lung carcinoma according to American Joint Committee on Cancer (AJCC) 7th edition or highly selected patients with oligo-metastatic disease amendable for thoracic radiotherapy with curative intent
3. Not undergoing radical surgical resection
4. Patients do not have prior radiotherapy to the thorax
5. Age ≥ 20 years
6. Karnofsky performance status (KPS) ≥ 60%.
7. Women of childbearing potential and male participants must practice adequate contraception
8. Patients must be able to comply with the study protocol and follow-up schedules and provide study-specific informed consent

Exclusion criteria:

1. Prior radiotherapy to thorax
2. Unable to receive assigned radiation dose due to normal lung constraint
3. Inability to attend full course of radiotherapy or follow-up visits
4. Presence of metastatic disease. Patients who present with oligo-metastatic disease where all metastases have been ablated (with surgery or radiotherapy) or in complete remission after systemic therapy are candidates if they are receiving radiotherapy to the thoracic disease with curative intent
5. Severe, active comorbidities which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and adverse events of the protocol, or limit compliance with study requirements, defined as follows:

   * Uncontrolled active infection requiring intravenous antibiotics at the time of registration
   * Transmural myocardial infarction ≤ 6 months prior to registration.
   * Unstable angina or congestive heart failure requiring hospitalization ≤ 6 months prior to registration.
   * Life-threatening uncontrolled clinically significant cardiac arrhythmias.
   * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects.
   * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration.
   * Uncontrolled psychiatric disorder.
6. Women of childbearing potential and male participants who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the radiation treatment involved in this study may be significantly teratogenic.
7. Pregnant or lactating women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2016-06; Primary Completion 2021-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
The pulmonary quality of life at 3 months post-radiotherapy | Change from Baseline Functional Assessment of Cancer Therapy-Lung Cancer Subscale at 3 months
  Functional Assessment of Cancer Therapy-Lung Cancer Subscale (FACT-LCS)

SECONDARY OUTCOMES:
Changes of pulmonary function test post-radiotherapy | At baseline, 3, 6, 12 months, and annually until year 5 post-radiotherapy
  Screening spirometry, diffusion capacity of lung for carbon monoxide
Patient reported outcome (Quality of Life questionnaire by Functional Assessment of Cancer Therapy) | At baseline, 1, 2, 3, 4, 6, 9 12 months post-radiotherapy
  Functional Assessment of Cancer Therapy-Lung
Patient reported outcome (Quality of Life questionnaire by EORTC Core) | At baseline, 1, 2, 3, 4, 6, 9 12 months post-radiotherapy
  EORTC Quality of Life-Core 30 questionnaire module
Patient reported outcome (Quality of Life questionnaire by EORTC Lung cancer) | At baseline, 1, 2, 3, 4, 6, 9 12 months post-radiotherapy
  EORTC Quality of Life questionnaire -Lung cancer 13
Acute toxicity | From date of radiotherapy until 90 days after radiotherapy starts
  Common Toxicity Criteria for Adverse Events version 4
Late toxicity | 90 days after radiotherapy starts until the date of death from any cause, up to 60 months
  Common Toxicity Criteria for Adverse Events version 4
Progression free survival | From date of enrollment until the date of first documented disease progression or date of death from any cause, whichever came first, assessed up to 60 months
  Number of participant without disease progression
Overall survival | From date of enrollment until the date of death from any cause, assessed up to 60 months
  Number of participant alive

OTHER OUTCOMES:
Serum biomarkers in association with radiation pneumonitis | At baseline, 1, 2, 3, 4, 6 months post-radiotherapy
  Tumor necrosis factor-alpha, Transforming growth factor-beta concentration measured by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Ming Hsu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided